CLINICAL TRIAL: NCT01352026
Title: Evaluation of Metformin Activity in Addition to Conventional Treatment of Grade II or III Pulmonary Arterial Hypertension (PAH)
Acronym: MetHTAP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Several therapeutic have been developed making more difficult the eligibility of patients - Recruitment of new centers wasn't possible due to competing trials
Sponsor: Nantes University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BRD10/6-V
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Metformin

ARMS (1):
- Metformin (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
Treatment of PAH includes exercise limitation, non specific agents (anticoagulants, diuretics and supplemental oxygen), pulmonary specific vasodilators and antiproliferative agents.

Recent data obtained by our group, within rat PAH models, showed that the antihyperglycemic drug metformin, used in France since 1959 in diabetic type II patients, significantly acts at the pulmonary arteries level.

According to these results, and knowing that metformin is a widely used drug, with a favorable safety profile, the investigators decided to set up a pilot study, in order to evaluate the activity of metformin in PAH treatment. In parallel, the investigators will focus on metformin mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged between 18 and 80
* Patients included will have pre-capillary PAH
* they have to be stable for more than 3 months
* Patient with a 6-minute walk test comparable over the last 3 months before inclusion
* Informed consent signed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05

PRIMARY OUTCOMES:
The primary objective of this study will be to demonstrate the improvement of walk test distance in patients with pulmonary arterial hypertension (PAH) treated by metformin.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Nantes, Nantes
  - CHU de Bordeaux, Pessac